CLINICAL TRIAL: NCT05917340
Title: Comparative Evaluation of Intensified Short Course Regimen and Standard Regimen for Adults TB Meningitis : an Open-label Randomized Controlled Trial
Brief Title: Intensified Short Course Regimen for TBM in Adults
Acronym: INSHORT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: All India Institute of Medical Sciences, Jodhpur (Other Government); Christian Medical College, Vellore, India (Other); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); North Eastern Indira Gandhi Regional Institute of Health ans Medical Sciences (Other Government); Madras Medical College (Other Government); Rural Development Trust Hospital (Other)
Responsible Party: Principal Investigator, Leeberk Raja Inbaraj, Scientist-E (Medical), Tuberculosis Research Centre, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIRT-IEC No:2023 003
Record Dates: First submitted 2023-06-08; First posted 2023-06-23 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Tuberculous Meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Rifampin; Moxifloxacin; Aspirin; Isoniazid; Pyrazinamide; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm- 1( Intervention arm with aspirin) (Experimental): Intensified with high dose rifampicin, moxifloxacin, aspirin and steroids in the initial two months.
  Interventions: Drug: High dose rifampicin (25mg/kg); Drug: Moxifloxacin 400mg; Drug: Aspirin 150 mg; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Steroid; Drug: Rifampicin
- Arm -2 (Intervention arm without aspirin) (Experimental): Intensified with high dose rifampicin, moxifloxacin and steroids in the initial two months.
  Interventions: Drug: High dose rifampicin (25mg/kg); Drug: Moxifloxacin 400mg; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Steroid; Drug: Rifampicin
- Arm -3 (Control) (Active Comparator): Regimen as per the current National Tuberculosis Elimination Program in India.
  Interventions: Drug: HRZE; Drug: HRE

INTERVENTIONS:
Drug: High dose rifampicin (25mg/kg) — Given for 2 months
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: Moxifloxacin 400mg — Given for 2 months
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: Aspirin 150 mg — Given for 2 months
  Arms: Arm- 1( Intervention arm with aspirin)
Drug: Isoniazid — Given for 6 months
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: Pyrazinamide — Given for 6 months
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: Steroid — Tapering dose of dexamethasone or prednisolone upto 8 weeks
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: Rifampicin — Standard dose for 4 months after the initial treatment with high dose
  Arms: Arm -2 (Intervention arm without aspirin); Arm- 1( Intervention arm with aspirin)
Drug: HRZE — 2 months
  Arms: Arm -3 (Control)
Drug: HRE — 7-10 months as per TB program guidelines
  Arms: Arm -3 (Control)

SUMMARY:
Tuberculous meningitis (TBM) is the most lethal form of extra pulmonary tuberculosis. This devastating disease kills almost a third of its sufferers and disables a significant proportion of the survivors. TBM poses one of the most difficult diagnostic and therapeutic challenges in modern clinical practice. High-quality robust clinical trials have made a considerable contribution to the treatment of pulmonary tuberculosis in the last four decades. However, evidence from such clinical trials is lacking in TBM and the treatment remains uncertain. There is a significant variation in the choice, dose and duration of drugs between countries, institutions and clinicians. Investigators propose a multi-centric open-label clinical trial to assess the efficacy of short-course anti-TB drugs with high dose rifampicin, and moxifloxacin along with conventional anti-TB drugs and adjuvant therapy with aspirin and corticosteroids. Controls will receive standard treatment as per national guidelines for TBM. The investigators also aim to assess the safety and tolerability of high-dose Rifampicin and Moxifloxacin and the Pharmacodynamics and Pharmacokinetics parameters of ATT (Rifampicin, INH, Moxifloxacin and Pyrazinamide) in CSF between the two groups

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for entry to the trial if ALL of the following conditions are satisfied

1. Adults (> 18 years) with or without HIV infection
2. Possible, probable or definite TBM according to Lancet consensus diagnostic criteria
3. Willing to give written informed consent
4. Is willing to have an HIV test.
5. Residing within 100 km of the study sites
6. Express willingness to attend the treatment centre for supervised treatment
7. Express willingness to adhere to the trial procedures and follow-up schedule.
8. Agrees to use effective barrier contraception during the period of the treatment in case of female participants

Exclusion Criteria:

Patients will not be eligible for the trial if they meet ANY of the following criteria

1. Known current/previous drug resistance to ATT (Rifampicin, INH, FQ)**
2. Concurrent or known diagnosis any other meningitis such as bacterial, viral, and fungal.
3. Currently having an uncontrolled cardiac arrhythmia or ECG abnormalities which are contradiction for the administration of moxifloxacin including prolonged QTc. QTc value define as >450 ms in males and >460 ms in females measured in lead II or V5 on a standard 12-lead ECG.
4. Has clinical icterus or hepatic impairment characterized by serum bilirubin level above the normal laboratory reference range with abnormal liver enzymes, or isolated alanine aminotransferase (ALT) and/ or aspartate aminotransferase (AST) levels above 5 times the upper limit of the normal laboratory reference range
5. Previous history of anti-TB treatment, If any, should not exceed one month in the past and not more than 7 days in the preceding one month.
6. pregnant or lactating women
7. rapid clinical deterioration or very sick and moribund during the screening process, renal failure, liver disease or any condition (social or medical) that in the opinion of the investigator would make trial participation unreliable or unsafe.
8. Has a known allergy to any of the drugs proposed to be used in the trial regimen

   * All participants with Rifampicin resistance will be excluded at baseline from the study. Participants with H, FQ and Z resistance identified from MGIT results done at baseline will be referred back to NTEP for appropriate management and their numbers will be compensated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 12 months
  Between two groups
Disability rate | 12 months
  Measured by Modified Rankin scale. A score of 0 to 2 will be considered as no disability and 3-5 will be considered as disability. 0 - no symptoms ; 5 - severe disability
Mortality rate | 12 months
Disability rate | 24 months
  Measured by Modified Rankin scale. A score of 0 to 2 will be considered as no disability and 3-5 will be considered as disability. 0 - no symptoms ; 5 - severe disability

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of high dose rifampicin, isoniazid, pyrazinamide and moxifloxacin (Subset of patients) | Between week 1 & 2
  Plasma Cmax, cerebrospinal fluid [CSF] Cmax, and plasma/CSF Cmax ratio
Time for maximal concentration of high dose rifampicin, isoniazid, pyrazinamide and moxifloxacin (Subset of patients) | Between week 1 & 2
  Plasma Tmax, cerebrospinal fluid [CSF] Tmax, and plasma/CSF Tmax ratio
Area Under the Curve (AUC) of high dose rifampicin, isoniazid, pyrazinamide and moxifloxacin (Subset of patients) | Between week 1 & 2
  Plasma Tmax, cerebrospinal fluid [CSF] Tmax, and plasma/CSF Tmax ratio
Grade 3 & 4 adverse events | 12 months
  Comparison of the number of participants who develop Grade 3 or Grade 4 adverse events (according to Division of AIDS (DAIDS) criteria) during treatment. Grade 1 - mild event ; Grade 2 - moderate event; Grade 3- severe event ;Grade 4 - potentially life-threatening
Grade 3 & 4 adverse events | 24 months
  Comparison of the number of participants who develop Grade 3 or Grade 4 adverse events (according to Division of AIDS (DAIDS) criteria) during treatment. Grade 1 - mild event ; Grade 2 - moderate event; Grade 3- severe event ;Grade 4 - potentially life-threatening
Quality of life (QoL) in both the arms and change in QoL during the follow up | 6,12 & 24 months
  Using WHO Short form -36 (SF-36), a questionnaire to assess health related outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- ICMR- National Institute for Research in Tuberculosis, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inbaraj LR, Manesh A, Ponnuraja C, Bhaskar A, Srinivasalu VA, Daniel BD. Comparative evaluation of intensified short course regimen and standard regimen for adults TB meningitis: a protocol for an open label, multi-center, parallel arms, randomized controlled superiority trial (INSHORT trial). Trials. 2024 May 2;25(1):294. doi: 10.1186/s13063-024-08133-6. PMID 38693583